CLINICAL TRIAL: NCT03349333
Title: A Multi-center, Single Arm, Safety and Efficacy Study of Pralatrexate With Vitamin B12 and Folic Acid Supplementation in Subjects With Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: A Single Arm Study Evaluating the Efficacy and Safety of Pralatrexate in Subjects With Relapsed or Refractory PTCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOT12-CN-301
Record Dates: First submitted 2016-07-26; First posted 2017-11-21 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-03

CONDITIONS: Refractory Peripheral T-Cell Lymphoma; Relapsed T-Cell Lymphoma
Keywords: FOT12-CN-301; PTCL (peripheral T-cell lymphoma); pralatrexate; vitamin B12; folic acid
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pralatrexate (Experimental): Vitamin B12 and folic acid will be taken concurrently with pralatrexate
  Interventions: Drug: pralatrexate; Dietary Supplement: Vitamin B12 and folic acid

INTERVENTIONS:
Drug: pralatrexate — Pralatrexate will be administered at a dose of 30 mg/m2/week for 6 weeks followed by 1 week of rest in a 7-week cycle. Pralatrexate administration occurs once a week during week 1 through week 6 of each cycle.
Dietary Supplement: Vitamin B12 and folic acid — The eligible subjects will receive vitamin supplementation at screening phase, at least 10 days prior to pralatrexate administration on cycle 1, dose 1. Vitamin supplementation will consist of vitamin B12 1 mg intramuscular (IM) q 8-10 weeks and folic acid 1.2mg by mouth (PO) once a day (QD). Once pralatrexate is permanently discontinued, vitamin supplementation should continue at least 1 month after the last pralatrexate dose, or longer at the discretion of the investigator.

SUMMARY:
This is a single arm, open-label, multi-center study designed to demonstrate the efficacy and safety of pralatrexate when administered concurrently with vitamin B12 and folic acid supplementation to patients with relapsed or refractory peripheral T-cell lymphoma(PTCL).

DETAILED DESCRIPTION:
The primary objective of this study is to confirm the objective response rate (ORR) among Chinese subjects with relapsed or refractory PTCL treated with pralatrexate together with concurrent vitamin B12 and folic acid supplementation

Primary endpoint is objective Response Rate by International Working Group Criteria

This study includes 3 phases: Screening, Treatment (pralatrexate) and Follow-up phases.

Screening Phase:

The screening phase will be up to 28 days duration (depending on availability of lab results).

Treatment (pralatrexate) Phase:

The start of study treatment (pralatrexate) is defined as the initiation of pralatrexate. Patients will attend the clinic weekly for 6 weeks of a 7-week cycle to receive pralatrexate, and will be examined by the treating physician. One cycle of pralatrexate therapy is 7 weeks in duration and consists of 6 weekly doses of pralatrexate administered via intravenous (IV) push over 3-5 minutes, followed by 1 week of rest.

Evaluation of response must be performed within 7 days prior to the projected first dose of cycle 2-4 and then within 7 days prior to the projected first dose of every even-numbered subsequent cycle (ie, prior to cycles 6, 8, etc.). Although radiological response assessments have been scheduled every 14 weeks, unscheduled radiological response assessments will be performed earlier if clinical progression is suspected.

Treatment with pralatrexate will continue until 24 months of administration, or until documented disease progression; unacceptable adverse event(s) indicating intolerance of the lowest study dose allowed (20 mg/m2/week); omission of 3 sequential doses of pralatrexate due to a treatment-related AE; 3-week lapse between pralatrexate doses; development of an AE, intercurrent illness, condition, or procedural complication that may interfere with the subject's participation; investigator's decision to withdraw the subject; subject withdraws consent; pregnancy of the subject; noncompliance with trial treatment or procedure requirements; or administrative reasons.

Follow-up phase:

All patients who received at least 1 dose of pralatrexate are to attend the Safety Follow-up Visit [30 (± 5) days after the last dose of pralatrexate] and the protocol defined procedures and evaluations will be performed.

After the Safety Follow-up Visit, Routine Follow-up Visits will be based on standard clinical care. All patients who received at least 1 dose of pralatrexate are to attend Routine Follow-up Visits, which will occur every 3 months (± 2 weeks) for determination of progression of disease, subsequent treatment initiation for T-cell lymphoma and survival after the Safety Follow-up Visit for a total duration of 24 months after the last dose of pralatrexate. The protocol-defined procedures/evaluations should be performed at each Routine Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has histologically/cytologically confirmed PTCL, using the World Health Organization (WHO) disease classification:

   1. PTCL not otherwise specified (NOS)
   2. Angioimmunoblastic T-cell lymphoma
   3. Anaplastic large cell lymphoma, ALK+
   4. Anaplastic large cell lymphoma, ALK-
   5. Extranodal NK/T-cell lymphoma - nasal type
   6. Enteropathy-associated T cell lymphoma
   7. Hepatosplenic T-cell lymphoma
   8. Subcutaneous panniculitis-like T-cell lymphoma
   9. Adult T-cell lymphoma/leukemia (human T-cell leukemia virus [HTLV] 1+)
   10. Aggressive NK-cell leukemia
   11. Transformed mycosis fungoides
2. Subject has to have documented progressive disease (PD) after at least 1 prior systemic treatment.
3. Subject may not have received an experimental drug or biologic as their only prior therapy. Subject must have clear PD after the last treatment received. Subject should have at least 1 biopsy from initial diagnosis or in the relapsed setting to confirm the diagnosis of PTCL. Subject must have recovered from the toxic effects of prior therapy.
4. Subjects with an enlarged lymph node or extranodal mass lesion clearly measurable in two perpendicular directions and greater than 1.5 cm maximum diameter on computed tomography performed within 14 days prior to study enrollment.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
6. At least 18 years of age.
7. Expected life expectancy ≥ 3 months.
8. Adequate hematological, hepatic, and renal function as defined by:

   * Absolute neutrophil count (ANC) ≥ 1000/uL (or 1*109/L), platelet count ≥ 100,000/uL (or 100*109/L) (at both screening and within 3 days prior to dosing on cycle 1, day 1)
   * Total bilirubin ≤ 1.5 mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X upper limit of normal (ULN) (AST/ALT < 5 X ULN if documented hepatic involvement with lymphoma)
   * Creatinine ≤ 1.5 mg/dL (or 132.6 µmol/L) or a calculated creatinine clearance ≥ 50 mL/min
9. Women of childbearing potential must have agreed to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 30 days after the last administration of pralatrexate and must have a negative serum pregnancy test within 14 days prior to the first day of study treatment. Subjects who are postmenopausal for at least 1 year (> 12 months since last menses) or are surgically sterilized did not require this test.
10. Men who are not surgically sterile must agree to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 90 days after the last administration of pralatrexate.
11. Subject gives written informed consent (IC).

Exclusion Criteria:

1. Subject has:

   1. Precursor T-cell lymphoma or leukemia
   2. T-cell prolymphocytic leukemia (T-PLL)
   3. T-cell large granular lymphocytic leukemia
   4. Mycosis fungoides, other than transformed mycosis fungoides
   5. Sézary syndrome
   6. Primary cutaneous CD30+ T-cell disorders: Lymphoid papulosis and primary cutaneous anaplastic large cell lymphoma
2. Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 5 years.
3. Congestive heart failure Class III/IV according to the New York Heart Association's Heart Failure guidelines.
4. Human immunodeficiency virus (HIV)-positive diagnosis.
5. Has, or history of, brain metastases or central nervous system (CNS) disease.
6. Active uncontrolled infection, underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of the subject to receive protocol treatment.
7. Has major surgery within 2 weeks of study entry.
8. Receipt of any conventional chemotherapy or radiation therapy (RT) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the course of the study.
9. Receipt of corticosteroids within 7 days of study treatment, unless subject has been taking a continuous systemic dose of no more than 10 mg/day or equivalent dose of prednisone, or a local or inhaled or intranasal administration at fixed doses for at least 1 month prior to study treatment and tumor shrinkage was not observed.
10. Use of any investigational drugs, biologics, or devices within 4 weeks prior to study treatment or planned use during the course of the study.
11. Receipt of anti-tumor antibody therapy within 100 days prior to study treatment.
12. History of allogeneic hematopoietic stem cell transplantation. Or subjects with a history of autologous hematopoietic stem cell transplantation within 100 days prior to study treatment.
13. Previous exposure to pralatrexate.
14. Subject is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria YU, Study Director — Mundipharma, China
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong X, Song Y, Huang H, Bai B, Zhang H, Ke X, Shi Y, Zhu J, Lu G, Liebscher S, Cai C. Pralatrexate in Chinese Patients with Relapsed or Refractory Peripheral T-cell Lymphoma: A Single-arm, Multicenter Study. Target Oncol. 2019 Apr;14(2):149-158. doi: 10.1007/s11523-019-00630-y. PMID 30904980

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the protocol, 85 patients are planned to enroll. However, 71 patients are treated in the real situation.
Period: Overall Study
Arm/Group | Pralatrexate
Started | 71
Completed | 0
Not Completed | 71
Not completed — Progression of Disease | 36
Not completed — Adverse Event | 11
Not completed — Other | 6
Not completed — Withdrawal by Subject | 5
Not completed — Conditions interfere with participation | 2
Not completed — Physician Decision | 2
Not completed — 3-week lapse between pralatrexate doses | 1
Not completed — Patients in treatment less than 24 month | 8

BASELINE CHARACTERISTICS:
Population: Safety population is 71
Groups:
- PTCL Subtype: Vitamin B12 and folic acid will be taken concurrently with pralatrexate
  pralatrexate: Pralatrexate will be administered at a dose of 30 mg/m2/week for 6 weeks followed by 1 week of rest in a 7-week cycle. Pralatrexate administration occurs once a week during week 1 through week 6 of each cycle.
  Vitamin B12 and folic acid: The eligible subjects will receive vitamin supplementation at screening phase, at least 10 days prior to pralatrexate administration on cycle 1, dose 1. Vitamin supplementation will consist of vitamin B12 1 mg intramuscular (IM) q 8-10 weeks and folic acid 1.2mg by mouth (PO) once a day (QD). Once pralatrexate is permanently discontinued, vitamin supplementation should continue at least 1 month after the last pralatrexate dose, or longer at the discretion of the investigator.
Arm/Group | PTCL Subtype
Number analyzed (Participants) | 71
Age, Customized [Mean (Standard Deviation); unit: years]
  Age(years) | 54.5 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 71
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 71
Baseline Characteristics [Count of Participants; unit: Participants]
  Subtype of PTCL from investigator: PTCL not otherwise specified (NOS) | 34
  Subtype of PTCL from investigator: Angioimmunoblastic T-cell lymphoma | 19
  Subtype of PTCL from investigator: Anaplastic large cell lymphoma, ALK+ | 2
  Subtype of PTCL from investigator: Anaplastic large cell lymphoma, ALK- | 7
  Subtype of PTCL from investigator: Extranodal NK/T-cell lymphoma - nasal type | 5
  Subtype of PTCL from investigator: Subcutaneous panniculitis-like T-cell lymphoma | 2
  Subtype of PTCL from investigator: Enteropathy-associated T cell lymphoma | 1
  Subtype of PTCL from investigator: Adult T-cell lymphoma/leukemia (human T-cell leuke | 1
  Subtype of PTCL from investigator: other | 0
  Subtype of PTCL from central review: PTCL not otherwise specified (NOS) | 34
  Subtype of PTCL from central review: Angioimmunoblastic T-cell lymphoma | 20
  Subtype of PTCL from central review: Anaplastic large cell lymphoma, ALK+ | 2
  Subtype of PTCL from central review: Anaplastic large cell lymphoma, ALK- | 6
  Subtype of PTCL from central review: Extranodal NK/T-cell lymphoma - nasal type | 5
  Subtype of PTCL from central review: Subcutaneous panniculitis-like T-cell lymphoma | 1
  Subtype of PTCL from central review: Enteropathy-associated T cell lymphoma | 1
  Subtype of PTCL from central review: Adult T-cell lymphoma/leukemia (human T-cell leuke | 1
  Subtype of PTCL from central review: other | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate(ORR) by International Working Group Criteria
Description: ORR defined as the percentage of subjects with CR, CRu or PR as Best Overall Response.Evaluation of response must be performed within 7 days prior to the projected first dose of cycle 2-4 and then within 7 days prior to the projected first dose of every even-numbered subsequent cycle (i.e. prior to cycles 6, 8, etc). Unscheduled radiological response assessments will be performed earlier if clinical progression is suspected.The primary analysis will be conducted once all subjects have completed cycle 5 treatment or discontinued before. Study treatment may continue per investigator judgment for a maximum of 24 months.
  Response will be assessed on the basis of clinical, radiological, and pathological criteria. Response will be assessed by independent central review and by the treating investigator. Central review assessors will be blinded to the response assessments by the treating investigator. The primary analysis will be based on response assessed by central review.
Time Frame: 2 years
Population: The primary analysis was based on the independent review data using the safety population, safety population is 71 for this study
Measure: Count of Participants; unit: Participants
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
Participants | 37

2. Secondary Outcome: Time to Response (TTR)
Description: Time to response was measured from first day of treatment to the first date of documented response.
Time Frame: 2 years
Population: The secondary analyses was performed using the safety population and repeated using the per-protocol population.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
months | 2.0947 (1.6590)

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was measured from treatment day 1 until event or censoring. An event was defined as the earliest of the following: death from any cause or disease progression. Subjects undergoing transplant or any other subsequent therapy prior to documentation of PD was censored at that time. Progression of disease deems as 1. 50% increase from nadir in the SPD of any previously identified abnormal node for PRs or nonresponders, 2.Appearance of any new lesion during or at the end of therapy as per IWC criteria.
Time Frame: 2 years
Population: The secondary analyses was performed using the safety population and repeated using the per-protocol population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
months | 4.76 [3.06 to 8.75]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from treatment day 1 until death or censoring.
Time Frame: 4 years
Population: The secondary analyses was performed using the safety population and repeated using the per-protocol population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
months | 18.00 [10.35 to NA] — This analysis is based on cut off data, there are no enough events to estimated upper limit of 95% CI of median OS.

5. Secondary Outcome: Duration of Responses
Description: Duration of response was measured from first day of documented response to disease progression or death, whatever comes first.
Time Frame: 4 years
Population: The secondary analyses was performed using the safety population and repeated using the per-protocol population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
months | 8.67 [3.32 to 14.13]

6. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events
Description: treatment emergent AE was scheduled to be collected during all subject visits, the data evaluated as clinical significant will be summarized and presented.
Time Frame: 4 years
Population: safety population
Measure: Number; unit: percentage of participants
Arm/Group | Pralatrexate
Number analyzed (Participants) | 71
percentage of participants | 98.6

7. Secondary Outcome: Area Under the Curve [AUC] for R-pralatrexate
Description: The PK endpoints was analysed using the PK population. The overall PK population is defined as all subjects who receive at least one dose of Investigational Medicinal Product (IMP) and have at least one primary PK parameter. Subjects with non-zero baseline concentrations of >5% of Cmax for either analyte (R-pralatrexate or S-pralatrexate) will be removed from the PK population.
Time Frame: Cycle 1 day1，Cycle 1 week 6(Pre-injection, end-injection, 30 and 60 minutes, and 3, 5, 8, 12, 18, 24, 48, and 72 hours post-end injection)
Population: Based on PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h*ng/ml
  Pralatrexate-R in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-R in Cycle 1 week 6（20mg/m2） | 2350.7402 (28.22)
  Pralatrexate-R in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 8
  Pralatrexate-R in Cycle 1 week 6（30mg/m2） | 3979.1069 (152.16)
  Pralatrexate-R in Cycle 1 day 1（30mg/m2）: number analyzed (Participants) | 14
  Pralatrexate-R in Cycle 1 day 1（30mg/m2） | 3586.2925 (43.70)

8. Secondary Outcome: Area Under the Curve [AUC] for S-pralatrexate
Description: as for outcome 7
Time Frame: Cycle 1 day 1, Cycle 1 week 6（Pre-injection, end-injection, 30 and 60 minutes, and 3, 5, 8, 12, 18, 24, 48, and 72 hours post-end injection）
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h*ng/ml
  Pralatrexate-S in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-S in Cycle 1 week 6（20mg/m2） | 1364.7686 (22.65)
  Pralatrexate-S in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 7
  Pralatrexate-S in Cycle 1 week 6（30mg/m2） | 2182.5078 (264.05)
  Pralatrexate-S in Cycle 1 day 1（30mg/m2）: number analyzed (Participants) | 7
  Pralatrexate-S in Cycle 1 day 1（30mg/m2） | 1674.8773 (38.32)

9. Secondary Outcome: Steady State Volume of Distribution [Vdss] for R-pralatrexate
Description: as for outcome 7
Time Frame: Cycle 1 day 1, Cycle 1 week6(Pre-injection, end-injection, 30 and 60 minutes, and 3, 5, 8, 12, 18, 24, 48, and 72 hours post-end injection)
Population: PK population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
L
  Pralatrexate-R Cycle 1 day1（30mg/m2） | 194.1589 (87.4028)
  Pralatrexate-R Cycle 1 week6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-R Cycle 1 week6（20mg/m2） | 344.2511 (109.8671)
  Pralatrexate-R Cycle 1 week6（30mg/m2）: number analyzed (Participants) | 9
  Pralatrexate-R Cycle 1 week6（30mg/m2） | 329.1892 (251.4938)

10. Secondary Outcome: Steady State Volume of Distribution [Vdss] for S-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
L
  Pralatrexate-S Cycle 1 Day 1 (30 mg/m2) | 517.1628 (292.2888)
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2): number analyzed (Participants) | 3
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2) | 1110.6541 (548.2687)
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2): number analyzed (Participants) | 9
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2) | 1680.6116 (2292.0216)

11. Secondary Outcome: Steady State Clearance [CLss] for R-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
L/h
  Pralatrexate-R Cycle 1 Day 1 (30 mg/m2) | 17.1914 (6.7903)
  Pralatrexate-R Cycle 1 Week 6 (20 mg/m2): number analyzed (Participants) | 3
  Pralatrexate-R Cycle 1 Week 6 (20 mg/m2) | 16.3789 (5.3859)
  Pralatrexate-R Cycle 1 Week 6 (30 mg/m2): number analyzed (Participants) | 9
  Pralatrexate-R Cycle 1 Week 6 (30 mg/m2) | 19.8406 (8.9265)

12. Secondary Outcome: Steady State Clearance [CLss] for S-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
L/h
  Pralatrexate-S Cycle 1 Day 1 (30 mg/m2) | 34.6341 (17.9816)
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2): number analyzed (Participants) | 3
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2) | 27.9794 (8.4317)
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2): number analyzed (Participants) | 9
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2) | 45.2022 (22.4576)

13. Secondary Outcome: Maximum Observed Plasma Concentration [Cmax] for R-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
ng/mL
  Pralatrexate-R in Cycle 1 day 1（30mg/m2） | 4649.6811 (83.74)
  Pralatrexate-R in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-R in Cycle 1 week 6（20mg/m2） | 2488.1502 (17.78)
  Pralatrexate-R in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 9
  Pralatrexate-R in Cycle 1 week 6（30mg/m2） | 5064.6667 (421.48)

14. Secondary Outcome: Maximum Observed Plasma Concentration [Cmax] for S-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
ng/mL
  Pralatrexate-S in Cycle 1 day 1（30mg/m2） | 3727.8582 (118.25)
  Pralatrexate-S in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-S in Cycle 1 week 6（20mg/m2） | 2325.5105 (24.22)
  Pralatrexate-S in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 9
  Pralatrexate-S in Cycle 1 week 6（30mg/m2） | 3439.9695 (697.55)

15. Secondary Outcome: Time of Cmax Observation [Tmax] for R-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h
  Pralatrexate-R in Cycle 1 day 1（30mg/m2） | 0.1000 [0.067 to 0.333]
  Pralatrexate-R in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-R in Cycle 1 week 6（20mg/m2） | 0.1000 [0.100 to 0.167]
  Pralatrexate-R in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 9
  Pralatrexate-R in Cycle 1 week 6（30mg/m2） | 0.1000 [0.067 to 0.250]

16. Secondary Outcome: Time of Cmax Observation [Tmax] for S-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h
  Pralatrexate-S in Cycle 1 day 1（30mg/m2） | 0.1000 [0.067 to 0.333]
  Pralatrexate-S in Cycle 1 week 6（20mg/m2）: number analyzed (Participants) | 3
  Pralatrexate-S in Cycle 1 week 6（20mg/m2） | 0.1000 [0.100 to 0.167]
  Pralatrexate-S in Cycle 1 week 6（30mg/m2）: number analyzed (Participants) | 9
  Pralatrexate-S in Cycle 1 week 6（30mg/m2） | 0.1000 [0.067 to 0.250]

17. Secondary Outcome: Terminal Phase Half-life [t1/2Z] for R-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h
  Pralatrexate-R Cycle 1 Day 1 (30 mg/m2): number analyzed (Participants) | 14
  Pralatrexate-R Cycle 1 Day 1 (30 mg/m2) | 8.5040 (3.4927)
  Pralatrexate-R Cycle 1 Week 6 (20 mg/m2): number analyzed (Participants) | 3
  Pralatrexate-R Cycle 1 Week 6 (20 mg/m2) | 14.6089 (0.1970)
  Pralatrexate-R Cycle 1 Week 6 (30 mg/m2): number analyzed (Participants) | 8
  Pralatrexate-R Cycle 1 Week 6 (30 mg/m2) | 11.8249 (4.3282)

18. Secondary Outcome: Terminal Phase Half-life [t1/2Z] for S-pralatrexate
Description: as for outcome 7
Time Frame: as for outcome 8
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Pralatrexate
Number analyzed (Participants) | 15
h
  Pralatrexate-S Cycle 1 Day 1 (30 mg/m2): number analyzed (Participants) | 7
  Pralatrexate-S Cycle 1 Day 1 (30 mg/m2) | 10.8634 (5.6517)
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2): number analyzed (Participants) | 3
  Pralatrexate-S Cycle 1 Week 6 (20 mg/m2) | 26.2505 (7.7381)
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2): number analyzed (Participants) | 7
  Pralatrexate-S Cycle 1 Week 6 (30 mg/m2) | 24.8987 (23.2607)

ADVERSE EVENTS:
Time Frame: AEs were recorded in the eCRF from the point at which the ICF was signed until 30 (± 5) days after the last dose of pralatrexate. This included new AEs that were reported in the 30 (± 5) days after the last dose of pralatrexate.
Arm/Group | Pralatrexate
All-Cause Mortality (participants affected / at risk) | 29/71
Serious Adverse Events (participants affected / at risk) | 35/71
Other Adverse Events (participants affected / at risk) | 70/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate (N=71)
Lung infection (Infections and infestations) | 7 (8)
Platelet count decreased (Investigations) | 10 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate (N=71)
Stomatitis (Gastrointestinal disorders) | 48 (101)
Neutropenia (Blood and lymphatic system disorders) | 22 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03349333/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03349333/SAP_001.pdf